CLINICAL TRIAL: NCT01615042
Title: Phase I Trial of High Dose Lenalidomide in Patients With Refractory/Relapsed Acute Leukemia as a Bridge to Bone Marrow Transplant
Brief Title: Phase I Study of Lenalidomide in Patients With Acute Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Mehrdad Abedi, MD (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Mehrdad Abedi, MD, Professor, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 318008; UCDCC#228 (Other: UC Davis); RV_AML_PI_0696 (Other: Celgene)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Acute Leukemia
Keywords: Acute Leukemia; Bone Marrow Transplant; High Dose Lenalidomide
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation/High Dose Lenalidomide (Experimental): Subjects are given a single dose of the drug while they are observed and tested for a period of time. If they do not exhibit any adverse side effects the dose is escalated, and a new group of subjects is then given a higher dose.
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Oral capsule, daily, 50mg-100mg, one cycle (21 days)
  Other Names: Revlimid

SUMMARY:
Lenalidomide is a drug that alters the immune system and it may also be directly toxic to tumor. Therefore, in theory, it may reduce or prevent the growth of cancer cells or directly kill them. We will be studying how lenalidomide can be used to decrease bone marrow blast cells in preparation for a bone transplant.

DETAILED DESCRIPTION:
We hypothesize that lenalidomide in high doses can be used to decrease bone marrow blast count in patients with relapsed or refractory acute myeloid leukemia in preparation for an allogeneic stem cell transplant with acceptable toxicities that are no worse than current cytotoxic chemotherapeutic agents. The known dose-limiting toxicity at 75 mg was excessive fatigue in a previous phase I trial which in this study may be irrelevant as all study participants will have an in-patient status.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Between 18 and 80 years of age at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Non-M3 Acute Myeloid Leukemia with the presence of residual disease in the bone marrow on day 14-28 post induction (or re-induction) chemotherapy. Day 14-28 residual disease is defined in this study as the presence of more than 10 % blasts in the marrow, presence of between 5-10% blasts cells that are not in cluster in hypocellular marrow is ambiguous and bone marrow biopsy should be repeated in 5-7 days.
* Patient should have an already identified sibling, matched unrelated donor or cord blood donor at the time of enrollment to this clinical trial.
* Eastern Cooperative Oncology Group (ECOG) performance status of equal or less than 3 at study entry (this patient population is typically admitted and is in the hospital)
* Laboratory test results within defined ranges
* Disease free of other malignancies beside the acute myeloid leukemia (AML) for greater than or equal to 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
* Females of childbearing potential (FCBP)must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International unit (mIU)/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide prescriptions must be filled within 7 days as required by RevAssist) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or breast feeding females (Lactating females must agree not to breast feed while taking lenalidomide).
* Patients younger than 50 years old, after first induction of chemotherapy, who are able to safely tolerate re-induction therapy with high dose chemotherapy are not eligible for this study.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Use of any other experimental drug or therapy within 14 days of baseline.
* Known hypersensitivity to thalidomide or lenalidomide (if applicable).
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known sero-positive for active viral infection with human immunodeficiency virus, hepatitis B virus or hepatitis C virus. Patients who are sero-positive because of hepatitis B virus vaccine are eligible.
* Patients who are not able to swallow the lenalidomide capsule as a whole are excluded from this study.
* Patients with impaired gastrointestinal absorption
* Symptomatic congestive heart failure
* Unstable angina pectoris or cardiac arrhythmia
* History of adrenal insufficiency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (measured by NCI Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0) | One Cycle (21 days)
  All patients who receive the study drug will be followed closely and evaluated for toxicity.
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL. Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE

SECONDARY OUTCOMES:
Rates of complete response (CR) and complete response without platelet recovery (CRi) | One Cycle (21 days)
  Patients will be assessed for the efficacy (CR or CRi) if they have received at least 7 continuous days of study drug.
Pharmacokinetics of high-dose lenalidomide cell activity. | At 0.25, 0.5, 1, 2, 3, 4, 6, 8, and 24 hours after dose on day 1, as well as before morning dosing on days 8, 15, and 21 during the clinical therapy
  Plasma concentrations of lenalidomide will be studied
Define the effects of lenalidomide on T and Natural Killer (NK) cell activity. | Baseline and at two weeks after therapy
  Blood samples will be drawn and will be tested for NK cell and T cell activity.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Abedi, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Comprehensive Cancer Center, Sacramento, California, United States

REFERENCES:
- See also: University of California Davis Comprehensive Cancer Center Website — http://www.ucdmc.ucdavis.edu/cancer/